CLINICAL TRIAL: NCT05691660
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Single and Multiple Dose Escalating Study of TAS3731 in Healthy Adults
Brief Title: A Study of TAS3731 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Taiho Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10074010
Record Dates: First submitted 2022-11-24; First posted 2023-01-20 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Healthy Adult Males

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single dose cohort (Experimental)
  Interventions: Drug: TAS3731 Dose1; Drug: Placebo
- Repeated dose cohort Once daily (QD) (Experimental)
  Interventions: Drug: TAS3731 Dose2; Drug: Placebo
- Repeated dose cohort Twice daily (BID) (Experimental)
  Interventions: Drug: TAS3731 Dose3; Drug: Placebo

INTERVENTIONS:
Drug: TAS3731 Dose1 — Oral administration,1 day,QD
  Arms: Single dose cohort
Drug: TAS3731 Dose2 — Oral administration,7 days,QD
  Arms: Repeated dose cohort Once daily (QD)
Drug: TAS3731 Dose3 — Oral administration,7 days,BID
  Arms: Repeated dose cohort Twice daily (BID)
Drug: Placebo — Oral administration, 1 day,QD
  Arms: Single dose cohort
Drug: Placebo — Oral administration, 7 days,QD
  Arms: Repeated dose cohort Once daily (QD)
Drug: Placebo — Oral administration, 7 days,BID
  Arms: Repeated dose cohort Twice daily (BID)

SUMMARY:
To evaluate the safety of single and repeated administration of TAS3731.

ELIGIBILITY:
Key Inclusion Criteria:

1. Healthy adult male subjects who provided written informed consent to participate in the study
2. Aged 18 years or older and younger than 40 years at the time of informed consent
3. Body weight of 50 kg or more at screening:
4. Body mass index of 18.5 or more and less than 25.0 (Japanese) or less than 30.0 kg/m2 (Caucasian)
5. Capable of oral intake.

Key Exclusion Criteria

1. Complications or history of diseases that may affect absorption, distribution, metabolism, or excretion of the investigational drug, such as hepatic/biliary tract disease, renal/urologic disease, or gastrointestinal disease. The stomach or small intestine has been resected.
2. The 12-lead electrocardiogram at the time of the screening test was judged by the investigator to be inadequate for this study.
3. Had any concurrent disease (including symptoms and signs; however, diseases that do not affect evaluations in the study such as asymptomatic pollinosis and wart are excluded)
4. The patient has the following complications or a history of the following.

   1. Had current or previous drug abuse (including use of illicit drugs) or alcoholism
   2. Had current or previous hypersensitivity or allergy to drugs
5. Suspected COVID-19 disease.

Ages: 18 Years to 39 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2023-01-17 (Actual); Primary Completion 2024-05-21 (Actual); Study Completion 2024-05-21 (Actual)

PRIMARY OUTCOMES:
The number and incidence rate of adverse events | Single dose cohort：Day 1 to 7, Repeated dose cohort：Day 1 to 16
The number and incidence rate of adverse drug reactions | Single dose cohort：Day 1 to 7, Repeated dose cohort：Day 1 to 16
Evaluation of Systolic and Diastolic blood pressure | Single dose cohort：Change from Baseline Systolic and Diastolic Blood Pressure at 7 days, Repeated dose cohort：Change from Baseline Systolic and Diastolic Blood Pressure at 16 days
Evaluation of pulse rate | Single dose cohort：Change from Baseline pulse rate at 7 days, Repeated dose cohort：Change from Baseline pulse rate at 16 days
Evaluation of body temperature | Single dose cohort：Change from Baseline body temperature at 7 days, Repeated dose cohort：Change from Baseline body temperature at 16 days
Number of participants with abnormal laboratory values | Single dose cohort：Change in number of participants with abnormal laboratory values between baseline and 7 days, Repeated dose cohort：Change in number of participants with abnormal laboratory values between baseline and 16 days
Evaluation of QT interval corrected for heart rate using Fridericia's formula(QTcF) interval | Single dose cohort：Change from Baseline QTcF interval at 7 days, Repeated dose cohort：Change from Baseline QTcF interval at 16 days
Evaluation of RR-interval | Single dose cohort：Change from Baseline Evaluation of RR-interval at 7 days, Repeated dose cohort：Change from Baseline Evaluation of RR-interval at 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Taiho Pharmaceutical Co., Ltd., Study Director — Taiho Pharmaceutical Co., Ltd.
Locations (1):
- A site selected by Taiho Pharmaceutical Co., Ltd., Tokyo, Japan

IPD SHARING:
Plan to Share IPD: No
Data will not be shared according to the Sponsor policy on data sharing. Taiho policy on data sharing may be found at https://www.taiho.co.jp/en/science/policy/clinical_trial_information_disclosure_policy/index.html.